CLINICAL TRIAL: NCT04742660
Title: The Effect of Administration of Glycyrrhizin During Induction Period on the Occurrence of Postoperative Nausea and Vomiting After Breast Surgery
Brief Title: The Effect of Glycyrrhizin on the Occurrence of Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Yea-Ji Lee, clinical assistant professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KUH
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2022-05

CONDITIONS: Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Glycyrrhizic Acid

STUDY DESIGN:
Intervention Model Description: The anticipants are administered either ramosetron+placebo or ramosetron+glycyrrhizin
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to allocated groups. Outcomes assessors are blinded to which group participants are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group R (Placebo Comparator): Participants are administered a dose of 0.3mg of ramosetron (conventional antiemetics) intravenously followed by continuous infusion of 120mL normal saline at a rate of 10mL/min.
  Interventions: Drug: Ammonium Glycyrrhizinate
- group G (Active Comparator): participants are administered a dose of 0.3mg of ramosetron followed by continuous infusion of mixture of 20mL glycyrrhizin and 100mL normal saline (total 120mL) at a rate of 10mL/min.
  Interventions: Drug: Ammonium Glycyrrhizinate

INTERVENTIONS:
Drug: Ammonium Glycyrrhizinate — In control group, we assess the incidence and severity of PONV when participants are aministered ramosetron and placebo. In intervention group, the outcomes are assessed as a result of administration of ramosetron and glycyrrhizin.
  Other Names: glycyrrhizin; gulucolin S

SUMMARY:
The investigators investigate the association between the administration of glycyrrhizin during induction of general anesthesia and the occurrence of postoperative nausea and vomiting (PONV) in patients undergo breast surgery

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is one of a common complication after general anesthesia with 30-50% of incidence, increased up to 80% in high risk group. The risk factors of PONV include women population, the previous history of PONV, motion sickness in usual life, non-smoker, exposure to inhalants, perioperative opioid and laparoscopic surgery. Women population is a strong risk factor of PONV. Although perioperative management of PONV based on a guideline has been done in a lot of medical centers worldwide, the incidence of PONV is still reported relatively high.

The main ingredient of Glycyrrhizin is liquorice which has been used as antispasmodics, antiemetics or treatment for gastric ulcer in oriental medicine. Utilizing these effects of liquorice, the investigators investigate whether the addition of glycyrrhzin to conventional antiemetics is effective to decrease the incidence of PONV and improvement of severity of PONV.

ELIGIBILITY:
Inclusion Criteria:

* participants scheduled to undergo breast surgery aged 20 and above

Exclusion Criteria:

* aldosteronism
* electrolyte imbalance
* myopathies
* drug addiction or suspected
* bowel disease
* allergy to drugs
* smoker
* taking any medications

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
the incidence of postoperative nausea and vomiting (PONV) | up to 24 hours after discharge from postanesthetic care unit (PACU)
  assessing the incidence of postoperative nausea and vomiting with ordinal scale (0=none, 1=nausea, 2=retching, 3= vomiting)

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hyop Kim, M.D. Ph.D, Study Director — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, Seoul-T'ǔkpyǒlshi, South Korea

IPD SHARING:
Plan to Share IPD: No